CLINICAL TRIAL: NCT01080612
Title: An Open-Label, Single-Dose, Randomized, Four-Way Crossover Study In Healthy Volunteers To Investigate The Pharmacokinetics Of Pregabalin Controlled Release Formulation Administered Following Various Caloric Intakes As Compared To The Immediate Release Formulation
Brief Title: A Study To Assess The Pharmacokinetics, Safety, And Tolerability Of A Pregabalin Controlled Release Formulation Administered Following Various Sized Caloric Meals As Compared To The Pregabalin Immediate Release Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A0081239
Record Dates: First submitted 2010-02-26; First posted 2010-03-04 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2010-07

CONDITIONS: Healthy
Keywords: pregabalin; pharmacokinetics; bioavailability
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 330 mg pregabalin controlled release: 400 to 500 calories (Experimental)
  Interventions: Drug: 330 mg pregabalin controlled release
- 330 mg pregabalin controlled release: 600 to 750 calories (Experimental)
  Interventions: Drug: 330 mg pregabalin controlled release
- 330 mg pregabalin controlled release: 800 to 1000 calories (Experimental)
  Interventions: Drug: 330 mg pregabalin controlled release
- 300 mg pregabalin immediate release (Other)
  Interventions: Drug: 300 mg pregabalin immediate release

INTERVENTIONS:
Drug: 330 mg pregabalin controlled release — A single dose of 330 mg controlled release tablet will be administered following a 400 to 500 calorie meal
  Arms: 330 mg pregabalin controlled release: 400 to 500 calories
Drug: 330 mg pregabalin controlled release — A single dose of 330 mg controlled release tablet will be administered following a 600 to 750 calorie meal
  Arms: 330 mg pregabalin controlled release: 600 to 750 calories
Drug: 330 mg pregabalin controlled release — A single dose of 330 mg controlled release tablet will be administered following an 800 to 1000 calorie meal
  Arms: 330 mg pregabalin controlled release: 800 to 1000 calories
Drug: 300 mg pregabalin immediate release — A single dose of 300 mg immediate release capsule will be administered in the fasted state
  Arms: 300 mg pregabalin immediate release

SUMMARY:
The purpose of this study is to (1) evaluate the effect of caloric intake on the pharmacokinetics of a single dose of a 330 mg pregabalin controlled release tablet relative to a 300 mg pregabalin immediate release capsule administered fasted and (2) determine the safety and tolerability of a single dose of a 330 mg pregabalin controlled release formulation administered following various sized caloric meals and the 300 mg pregabalin immediate release capsule administered fasted.

DETAILED DESCRIPTION:
To assess the single dose pharmacokinetics, safety, and tolerability of pregabalin controlled release formulation following various sized caloric meals relative to the immediate release formulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or females
* Between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2

Exclusion Criteria:

* Illicit drug use
* Pregnant or nursing females
* Females of childbearing potential who are unwilling or unable to use an acceptable method of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Pregabalin area under the curve (AUC) from time of study drug administration to the last quantifiable plasma concentration (AUClast) and to infinity (AUCinf) | 3 days

SECONDARY OUTCOMES:
Adverse events, vital signs, and clinical safety laboratories. | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Chew ML, Plotka A, Alvey CW, Pitman VW, Alebic-Kolbah T, Scavone JM, Bockbrader HN. Pharmacokinetics of pregabalin controlled-release in healthy volunteers: effect of food in five single-dose, randomized, clinical pharmacology studies. Clin Drug Investig. 2014 Sep;34(9):617-26. doi: 10.1007/s40261-014-0211-4. PMID 25078976
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081239&StudyName=A%20Study%20To%20Assess%20The%20Pharmacokinetics%2C%20Safety%2C%20And%20Tolerability%20Of%20A%20Pregabalin%20Controlled%20Release%20Formulation%20Administered%20Following%20V